CLINICAL TRIAL: NCT04445207
Title: Experimental Expanded Access Treatment With Convalescent Plasma for the Treatment of Patients With COVID-19
Status: No longer available | Type: Expanded Access
Sponsor: Jonathan Gerber (Other)
Responsible Party: Sponsor-Investigator, Jonathan Gerber, Associate Professor, University of Massachusetts, Worcester
Organization: University of Massachusetts, Worcester (Other)
Other Study IDs: H000020420
Record Dates: First submitted 2020-06-20; First posted 2020-06-24 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: COVID; Sars-CoV2; Corona Virus Infection
Keywords: COVID-19; Coronavirus; Sars-CoV2
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Biological: Convalescent Plasma — One to two 200 mL units of Convalescent plasma per infusion, up to 6 total units within a 3-week period.

SUMMARY:
The purpose of this program is to see if giving convalescent plasma to individuals who test positive for COVID-19 may reduce their symptoms and help minimize complications from the illness.

DETAILED DESCRIPTION:
As individuals are exposed to pathogens, the body's immune system works to create antibodies toward those pathogens. These antibodies can be found in the plasma portion of the blood. This plasma is referred to as "Convalescent plasma" and contains these infection fighting antibodies. Through a blood donation, this convalescent plasma is collected from a recovered person and transfused to a sick patient who is still fighting the same virus. This protocol will make convalescent COVID-19 plasma available to individuals who meet the eligibility criteria described.

ELIGIBILITY:
Inclusion Criteria:

* At least 12 years of age
* Covid-19 Convalescent Plasma (CCP) treatment is in line with the patient's current goals of care (i.e. recipient cannot be DNI status)
* Laboratory confirmed diagnosis of infection with SARS-CoV-2 that is severe or life threatening OR the individual is judged by the treating provider to be at a high risk of progression to severe or life-threatening disease.
* Severe COVID-19 is defined by one or more of the following:

  1. Dyspnea
  2. Respiratory frequency ≥ 30/min
  3. Blood oxygen saturation ≤ 93%
  4. Partial pressure of arterial oxygen to fraction of inspired oxygen ratio < 300
  5. Lung infiltrates > 50% within 24-48 hours
* Life-threatening COVID-19 is defined as one or more of the following:

  1. Respiratory failure
  2. Septic shock
  3. Multiple organ dysfunction or failure

Exclusion Criteria:

* History of prior life-threatening reactions to transfusion of blood products
* Not receiving other therapies that would preclude plasma transfusion

Min Age: 12 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Gerber, MD, Principal Investigator — UMASS MEDICAL SCHOOL
Locations (1):
- UMass Medical School, Worcester, Massachusetts, United States